CLINICAL TRIAL: NCT01373450
Title: Evaluation of the Glucoregulatory Effects of GLP-1 Receptor Activation in Patients With Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Glucoregulatory Effects of Glucagon-like Peptide-1 Receptor (GLP-1 Receptor) Activation in Participants With Type 2 Diabetes Mellitus (MK-0000-222)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000-222
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Oxyntomodulin; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- OXM → Lg-0.6 → Pbo → Lg-1.2 (Experimental): Participants received Oxyntomodulin 3.0 pmol/kg/min in the first, Liraglutide 0.6 mg in the second, Placebo in the third, and Liraglutide 1.2 mg in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide
- Lg-0.6 → Pbo → OXM → Pbo (Experimental): Participants received Liraglutide 0.6 mg in the first, Placebo in the second, Oxyntomodulin 3.0 pmol/kg/min in the third, and Placebo in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide
- Pbo → OXM → Lg-0.6 → Pbo (Experimental): Participants received Placebo in the first, Oxyntomodulin 3.0 pmol/kg/min in the second, Liraglutide 0.6 mg in the third, and Placebo in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide
- Lg-0.6 → OXM → Pbo → Lg-1.2 (Experimental): Participants received Liraglutide 0.6 mg in the first, Oxyntomodulin 3.0 pmol/kg/min in the second, Placebo in the third and Liraglutide 1.2 mg in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Liraglutide 1.2 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide
- OXM → Pbo → Lg-0.6 → Pbo (Experimental): Participants received Oxyntomodulin 3.0 pmol/kg/min in the first; Placebo in the second, Liraglutide 0.6 mg in the third, and Placebo in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide
- Pbo → Lg-0.6 → OXM → Lg-1.2 (Experimental): Participants received Placebo in the first, Liraglutide 0.6 mg in the second, Oxyntomodulin 3.0 pmol/kg/min in the third, and Liraglutide 1.2 mg in the fourth period
  Interventions: Drug: Oxyntomodulin; Drug: Liraglutide 0.6 mg; Drug: Liraglutide 1.2 mg; Drug: Placebo for Oxyntomodulin; Drug: Placebo for Liraglutide

INTERVENTIONS:
Drug: Oxyntomodulin — 3.0 pmol/kg/min as an intravenous (IV) infusion in the morning of the day of graded glucose infusion (GGI) (Day 1)
Drug: Liraglutide 0.6 mg — Single subcutaneous dose in the evening of the day before the GGI (Day-1)
  Other Names: Victoza®
Drug: Liraglutide 1.2 mg — Single subcutaneous dose in the evening of the day before the GGI (Day-1)
  Other Names: Victoza®
  Arms: Lg-0.6 → OXM → Pbo → Lg-1.2; Pbo → Lg-0.6 → OXM → Lg-1.2
Drug: Placebo for Oxyntomodulin — IV infusion in the morning of the day of GGI (Day 1)
Drug: Placebo for Liraglutide — Single subcutaneous dose in the evening of the day before the GGI (Day-1)

SUMMARY:
This was a four-period crossover study to assess the glycemic effects of a single dose of oxyntomodulin (OXM) on the glucose levels in participants with Type 2 diabetes mellitus (T2DM). Participants were randomly assigned to 1 of 6 treatment sequences consisting of 4 treatment periods, with a 7-day wash-out between each treatment period. The primary hypothesis was that during graded glucose infusion (GGI) oxyntomodulin (OXM) is neutral or better than placebo (Pbo) at lowering ambient plasma glucose levels, and at significantly enhancing insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≤38.0 kg/m^2
* Have a clinical diagnosis of Type 2 diabetes mellitus
* Have a glycated hemoglobin (HbA1C) at screening ≤9.0%; fasting plasma glucose should not exceed 300 mg/dL (16.8 mmol/L)
* Judged to be in good health

Exclusion Criteria:

* Have a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Have a history of stroke, chronic seizures, major neurological disorder, clinically significant endocrine, cardiovascular, hematological, hepatic, renal, respiratory, or genitourinary abnormalities or diseases
* Have untreated hypertension with blood pressure of >160/95 mmHg
* Have a history of neoplastic disease within the past 5 years
* Have a history of hypersensitivity to OXM, liraglutide, insulin or Haemaccel®
* Unable or unwilling to comply with restrictions around concomitant medications
* Consume excessive amounts of alcohol, coffee, tea, cola, or other caffeinated beverages daily
* Have had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks
* Have a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Currently a regular user (including use of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months
* Are unwilling or unable to consume the standardized meals during the study and/or is on a carbohydrate restricted diet (i.e., a diet <100 grams per day of carbohydrate)

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

REFERENCES:
- [Derived] Shankar SS, Shankar RR, Mixson LA, Miller DL, Pramanik B, O'Dowd AK, Williams DM, Frederick CB, Beals CR, Stoch SA, Steinberg HO, Kelley DE. Native Oxyntomodulin Has Significant Glucoregulatory Effects Independent of Weight Loss in Obese Humans With and Without Type 2 Diabetes. Diabetes. 2018 Jun;67(6):1105-1112. doi: 10.2337/db17-1331. Epub 2018 Mar 15. PMID 29545266
- [Derived] Shankar SS, Shankar RR, Mixson LA, Miller DL, Chung C, Cilissen C, Beals CR, Stoch SA, Steinberg HO, Kelley DE. Linearity of beta-cell response across the metabolic spectrum and to pharmacology: insights from a graded glucose infusion-based investigation series. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E865-73. doi: 10.1152/ajpendo.00527.2015. Epub 2016 Apr 12. PMID 27072496

RESULTS

PARTICIPANT FLOW:
Groups:
- OXM --> Lg-0.6--> Pbo--> Lg-1.2: Participants received Oxyntomodulin (OXM) 3.0 pmol/kg/min in the first, Liraglutide (Lg) 0.6 mg in the second, Placebo (Pbo) in the third, and Liraglutide 1.2 mg in the fourth period
- Lg-0.6 mg--> Pbo--> OXM--> Pbo: Participants received Liraglutide 0.6 mg in the first, Placebo in the second, Oxyntomodulin 3.0 pmol/kg/min in the third, and Placebo in the fourth period
- Pbo--> OXM--> Lg-0.6-->Pbo: Participants received Placebo in the first, Oxyntomodulin 3.0 pmol/kg/min in the second, Liraglutide 0.6 mg in the third, and Placebo in the fourth period
- Lg-0.6--> OXM--> Pbo--> Lg-1.2: Participants received Liraglutide 0.6 mg in the first, Oxyntomodulin 3.0 pmol/kg/min in the second, Placebo in the third and Liraglutide 1.2 mg in the fourth period
- OXM--> Pbo--> Lg-0.6--> Pbo: Participants received Oxyntomodulin 3.0 pmol/kg/min in the first; Placebo in the second, Liraglutide 0.6 mg in the third, and Placebo in the fourth period
- Pbo--> Lg-0.6--> OXM--> Lg-1.2: Participants received Placebo in the first, Liraglutide 0.6 mg in the second, Oxyntomodulin 3.0 pmol/kg/min in the third, and Liraglutide 1.2 mg in the fourth period
Period: Crossover Period 1
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 7 Day Wash-out
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Period 2
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 7 Day Wash-out
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Period 3
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 7 Day Wash-out
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Period 4
Arm/Group | OXM --> Lg-0.6--> Pbo--> Lg-1.2 | Lg-0.6 mg--> Pbo--> OXM--> Pbo | Pbo--> OXM--> Lg-0.6-->Pbo | Lg-0.6--> OXM--> Pbo--> Lg-1.2 | OXM--> Pbo--> Lg-0.6--> Pbo | Pbo--> Lg-0.6--> OXM--> Lg-1.2
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Treated Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-weighted Average of Glucose Measured by Area Under the Curve (AUC) After a Single Dose of Oxyntomodulin (OXM)
Description: Participants received on Day (-1) an overnight intravenous (IV) infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single dose of liraglutide (Lg) or placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 OXM or placebo for OXM, accompanied by up to 160 minutes of graded glucose infusion (GGI). During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting approximately 40 minutes. Glucose levels were measured from blood collected at baseline and during GGI at the following minutes: 0, 20, 40, 60, 80, 100, 120, 140, 160 and 165 in order to calculate the time-weighted average change from baseline in glucose AUC from 0-160 minutes.
Time Frame: Baseline and during GGI at time points 0, 20, 40, 60, 80, 100, 120, 140, 160 and 165 minutes
Population: Participants treated with Oxyntomodulin or placebo. Six participants were treated for two periods with placebo, resulting in placebo n = 18. Participants treated with Liraglutide were not analyzed for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Groups:
- Oxyntomodulin: Oxyntomodulin 3.0 pmol/kg/min IV infusion
- Placebo: Placebo for Oxyntomodulin IV infusion and Placebo for Liraglutide subcutaneous
Arm/Group | Oxyntomodulin | Placebo
Number analyzed (Participants) | 12 | 18
mg/dL | 106.3 (23.03) | 122.6 (35.29)
Statistical Analysis 1: Comparison: Oxyntomodulin vs Placebo; Test type: Superiority or Other; p = 0.024, t-test, 1 sided; Geometric Mean Ratio = 0.87, 90% CI 2-sided [0.77 to 0.98]

2. Primary Outcome: Change From Baseline in Maximum Ambient Glucose Concentration (Gmax) After a Single Dose of OXM
Description: Participants received on Day (-1) an overnight IV infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single dose of Lg or placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 OXM or placebo for OXM, accompanied by up to 160 minutes of GGI. During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting approximately 40 minutes. Glucose levels were measured from blood collected at baseline and during GGI to determine the maximum ambient glucose concentration above baseline.
Time Frame: Baseline and up to 160 minutes after start of GGI
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oxyntomodulin | Placebo
Number analyzed (Participants) | 12 | 18
mg/dL | 211.0 (63.00) | 272.9 (50.05)
Statistical Analysis 1: Comparison: Oxyntomodulin vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 1 sided; Geometric Mean Ratio = 0.77, 90% CI 2-sided [0.66 to 0.90]

3. Primary Outcome: Change From Baseline in Beta Cell Sensitivity to Glucose (Φ) After a Single Dose of OXM
Description: Beta cell sensitivity measures the ability to mount an insulin secretory response relative to the level of ambient plasma glucose. Participants received on Day (-1) an overnight IV infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single dose of Lg or placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 a single dose of OXM or placebo for OXM, accompanied by up to 160 minutes of GGI. During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting 40 minutes. Glucose (G), insulin and C-peptide levels were measured from blood collected at baseline and during GGI, with the decay in C-peptide concentration used to indirectly estimate the Insulin Secretion Rate (ISR). Beta Cell Sensitivity (Φ) was determined from the regression of the ISR on ambient plasma glucose (G).
Time Frame: Baseline and up to160 minutes after start of GGI
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: ISR (ng/mL) / Glucose (mg/dL)
Arm/Group | Oxyntomodulin | Placebo
Number analyzed (Participants) | 12 | 18
ISR (ng/mL) / Glucose (mg/dL) | 0.019 (0.010) [lower limit 0.013] | 0.006 (0.003)
Statistical Analysis 1: Comparison: Oxyntomodulin vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Least Square Mean Difference = 0.014, 90% CI 2-sided [0.008 to 0.019]

4. Secondary Outcome: Change From Baseline in Insulinotrophic Effect (ISR/G) at the Highest Glucose Infusion Rate After Two Periods of Placebo Treatment
Description: The reproducibility of insulinotrophic effects was compared after two separate placebo treatment periods within the same treatment sequence. Participants received on Day (-1) an overnight IV infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single subcutaneous dose of placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 placebo for OXM, accompanied by up to 160 minutes of GGI. During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting approximately 40 minutes. Over these two treatment periods glucose (G), insulin and C-peptide levels were measured from blood collected at the highest glucose infusion rate; with the decay in C-peptide concentration used to indirectly estimate the Insulin Secretion Rate (ISR), and hence to determine the insulinotrophic effect, ISR/G.
Time Frame: Baseline and 160 minutes after start of GGI at each placebo treatment period
Population: Participants within the same treatment sequence who were treated with Placebo in two separate treatment periods. Participants treated with Oxyntomodulin or Liraglutide were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ISR (ng/mg) / Glucose (mg/dL)
Groups:
- Placebo Period 1; Placebo Period 2: Placebo for Oxyntomodulin IV infusion and Placebo for Liraglutide subcutaneous
Arm/Group | Placebo Period 1 | Placebo Period 2
Number analyzed (Participants) | 6 | 6
ISR (ng/mg) / Glucose (mg/dL) | 0.0075 (0.0031) | 0.0070 (0.0027)
Statistical Analysis 1: Comparison: Placebo Period 1 vs Placebo Period 2; Test type: Superiority or Other; Intraclass Correlation Coefficient = 0.92, 90% CI 2-sided [0.72 to 0.98]

5. Secondary Outcome: Change From Baseline in Gmax After Single Doses of 0.6 mg Lg, or 1.2 mg Lg, Compared With Single Doses of Placebo or OXM
Description: Participants received on Day (-1) an overnight IV infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single dose of Lg or placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 a single dose of OXM or placebo for OXM, accompanied by up to 160 minutes of GGI. During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting approximately 40 minutes. Glucose levels were measured from blood collected at baseline and during GGI to determine the maximum ambient glucose concentration above baseline.
Time Frame: Baseline and up to 160 minutes after start of GGI
Population: All treated participants. Six participants were treated for two periods with placebo, resulting in a placebo n = 18.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Groups:
- Liraglutide 0.6 mg: Liraglutide 0.6 mg subcutaneous
- Liraglutide 1.2 mg: Liraglutide 1.2 mg subcutaneous
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Oxyntomodulin | Placebo
Number analyzed (Participants) | 12 | 6 | 12 | 18
mg/dL | 209.7 (66.08) | 157.9 (93.36) | 211.0 (63.00) | 272.9 (50.05)
Statistical Analysis 1: Comparison: Liraglutide 0.6 mg vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 1 sided; Geometric Mean Ratio = 0.77, 90% CI 2-sided [0.66 to 0.90]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Geometric Mean Ratio = 0.58, 90% CI 2-sided [0.45 to 0.74]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Oxyntomodulin; Test type: Superiority or Other; p = 0.473, t-test, 1 sided; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.85 to 1.16]
Statistical Analysis 4: Comparison: Liraglutide 1.2 mg vs Oxyntomodulin; Test type: Superiority or Other; p = 0.049, t-test, 1 sided; Geometric Mean Ratio = 0.75, 90% CI 2-sided [0.56 to 1.00]

6. Secondary Outcome: Change From Baseline in Insulinotrophic Effect (ISR/G) After Single Doses of 0.6 mg Lg, or 1.2 mg Lg, Compared With Single Doses of Placebo or OXM
Description: Participants received on Day (-1) an overnight IV infusion of insulin titrated to achieve baseline fasting plasma glucose on Day 1 of between 90 and 130 mg/dL. Participants also received on Day (-1) a single dose of Lg or placebo for Lg, after which insulin infusion was discontinued. Following overnight fast, participants received on Day 1 a single dose of OXM or placebo for OXM, accompanied by up to 160 minutes of GGI. During GGI glucose (20% D/W) was gradually infused at rates of 2,4,6 and 10 mg/kg/min, with each rate lasting approximately 40 minutes. Glucose (G), insulin and C-peptide levels were measured from blood collected at baseline and during GGI; with the decay in C-peptide concentration used to indirectly estimate the Insulin Secretion Rate (ISR) and hence determine ISR/G.
Time Frame: Baseline and up to 160 minutes after start of GGI
Population: All treated participants. Six participants were treated for two periods with placebo, resulting in placebo n = 18.
Measure: Least Squares Mean (Standard Deviation); unit: ISR (ng/min) / Glucose (mg/dL)
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Oxyntomodulin | Placebo
Number analyzed (Participants) | 12 | 6 | 12 | 18
ISR (ng/min) / Glucose (mg/dL) | 0.026 (0.015) | 0.035 (0.018) | 0.019 (0.010) | 0.006 (0.003)
Statistical Analysis 1: Comparison: Liraglutide 0.6 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Least Square Mean Difference = 0.021, 90% CI 2-sided [0.015 to 0.026]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Least Square Mean Difference = 0.030, 90% CI 2-sided [0.021 to 0.038]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Oxyntomodulin; Test type: Superiority or Other; p = 0.0163, t-test, 1 sided; Least Square Mean Difference = 0.007, 90% CI 2-sided [0.002 to 0.012]
Statistical Analysis 4: Comparison: Liraglutide 1.2 mg vs Oxyntomodulin; Test type: Superiority or Other; p = 0.0056, t-test, 1 sided; Least Square Mean Difference = 0.016, 90% CI 2-sided [0.006 to 0.026]

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study medication
Arm/Group | Oxyntomodulin | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 7/12 | 1/6 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxyntomodulin (N=12) | Liraglutide 0.6 mg (N=12) | Liraglutide 1.2 mg (N=6) | Placebo (N=12)
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Catheter Site Pain (General disorders) | 0 | 0 | 1 | 1
Catheter Site Related Reaction (General disorders) | 1 | 0 | 0 | 2
Fatigue (General disorders) | 2 | 3 | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.